CLINICAL TRIAL: NCT00005857
Title: Randomized Phase II Trial of Herceptin (NSC 688097) and Weekly Docetaxel (NSC 628503) in Androgen-Independent (Horomone Refractory) Adenocarcinoma of the Prostate (CaP)
Brief Title: Trastuzumab and Docetaxel in Treating Patients Who Have Metastatic Prostate Cancer That Is Refractory to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 99118; U01CA063265 (NIH); P30CA033572 (NIH); CHNMC-PHII-19; CHNMC-IRB-99118; NCI-T98-0090; CDR0000067884 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-06-02; First posted 2003-08-29 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Trastuzumab; Docetaxel

INTERVENTIONS:
Biological: trastuzumab
Drug: docetaxel

SUMMARY:
RATIONALE: Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to compare the effectiveness of trastuzumab alone and in combination with docetaxel in treating patients who have metastatic prostate cancer that is refractory to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy and toxicity of docetaxel (arm I) vs trastuzumab (Herceptin) (arm II), followed by a combination of docetaxel and trastuzumab in patients with androgen-independent or hormone-refractory metastatic, Her2/neu-positive prostate cancer. (Arm I closed to accrual effective 07/30/2001.)

OUTLINE: This is a multicenter study.

* Arm I: Patients receive docetaxel IV over 1 hour weekly for 6 weeks. Treatment continues every 8 weeks for at least 2 courses in the absence of unacceptable toxicity. (Arm I closed to accrual effective 07/30/2001. Arm I patients crossover to arm II.)
* Arm II: Patients receive trastuzumab (Herceptin) IV over 30-90 minutes weekly for 8 weeks. Treatment continues every 8 weeks for at least 2 courses in the absence of unacceptable toxicity.

Patients with progressive or stable disease after 2 courses of single-agent therapy receive docetaxel IV over 1 hour on day 1 of each week for 6 consecutive weeks and trastuzumab IV over 30-90 minutes on day 1 of each week for 8 consecutive weeks. Treatment continues every 8 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients with complete or partial response to single-agent therapy continue on that therapy until experiencing progressive or stable disease. The patients then proceed to combination therapy.

Patients are followed until death.

PROJECTED ACCRUAL: A total of 108-160 patients (54-80 per treatment arm) will be accrued for this study. (Arm I closed to accrual effective 07/30/2001.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV prostate cancer (any T, any N, M1, any G; D3)
* Clinical evidence of metastatic disease in bone or soft tissue
* Her2/neu-positive (2+ and 3+) by immunochemistry or fluorescent in situ hybridization
* Androgen-independent

  * Serum PSA at least 10 ng/mL that has risen on 3 successive evaluations after prior hormonal therapy
  * At least 1 month since prior antiandrogen therapy (e.g., flutamide, bicalutamide, or nilutamide) and rising PSA levels with 1 of the 2 rising PSA levels, measured at least 2 weeks apart, after antiandrogen withdrawal
* Bone only disease and elevated PSA alone allowed
* LHRH analog therapy must continue in patients who have not had prior orchiectomy and have castrate levels of testosterone

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm3
* Absolute granulocyte count at least 1,800/mm3
* Platelet count at least lower limit of normal (LLN)

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.6 mg/dL
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* Ejection fraction more than 50% or more than LLN by MUGA scan or 2-D echocardiogram
* No symptomatic coronary artery disease
* No active ischemia on EKG

Other:

* Fertile patients must use effective contraception
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* No more than one prior nonanthracycline chemotherapy regimen (including suramin)

Endocrine therapy:

* See Disease Characteristics
* No concurrent corticosteroids as antiemetic

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* At least 3 months since prior strontium chloride Sr 89 and recovered
* No concurrent radiotherapy to measurable lesions

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (4):
- United States (4):
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - St. Elizabeth's Medical Center of Boston, Brighton, Massachusetts

REFERENCES:
- [Result] Lara PN Jr, Chee KG, Longmate J, Ruel C, Meyers FJ, Gray CR, Edwards RG, Gumerlock PH, Twardowski P, Doroshow JH, Gandara DR. Trastuzumab plus docetaxel in HER-2/neu-positive prostate carcinoma: final results from the California Cancer Consortium Screening and Phase II Trial. Cancer. 2004 May 15;100(10):2125-31. doi: 10.1002/cncr.20228. PMID 15139054